CLINICAL TRIAL: NCT05039255
Title: Acute Effects of Self-correcting Movement on the Balance and Spine of Patients With Scoliosis. Observational Clinical Study
Brief Title: Acute Effects of Self-correcting Movement on the Balance and Spine of Patients With Scoliosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: UPavia
Record Dates: First submitted 2021-09-07; First posted 2021-09-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Scoliosis Idiopathic
Keywords: Scoliosis; self elongation movement; balance; spine curves
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the acute effects of the self-elongation movement on the balance of patients (aged 8-16 years) suffering from adolescent idiopathic scoliosis,

DETAILED DESCRIPTION:
Recruitment will be carried out by the physician during the scheduled follow-up. The participant and both parents, or the legal guardian, will receive information on the purpose and methods of this study. The informed consent of both parents, or the legal guardian, and of the minor will be requested.

Balance data (oscillations, sway area) will be collected by letting participants get on a stabilometric platform and placing their feet on the landmarks; position will not change for the duration of the assessments.

At the same time, the modification of the amplitude of the scoliotic curves will be evaluated with the use of the Spine 3D (medical class system) which uses micro-pulse laser technology to make a three-dimensional reconstruction of the spine.

Three 10-seconds assessments will be made. In the first the subject will reproduce the position hold for the scheduled radiography and an acquisition will be performed with the Spine3D. The obtained image will be compared with the radiographic one to improve the accuracy of the next evaluations. During the last two acquisitions, the stabilometric platform and the 3D Spine will be used simultaneously and the data for the study will be collected. The second acquisition will be performed in a physiological position and the third in self-lengthening, a position used in most of the rehabilitation methods for scoliosis. The full evaluation will take approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic scoliosis, carried out by the Physician with the Adams test and the scoliometer;
* age between 8 and 16 years, both sexes;
* ability to perform the self-elongation movement;
* amplitude of the major scoliotic curve <40 degrees Cobb;
* scheduled annual follow-up which requires a radiograph.

Exclusion Criteria:

* secondary scoliosis;
* obesity;
* orthopedic pathologies that modify the plantar supports;
* pathologies that modify balance (neurological and / or vestibular);
* inability to understand and sign informed consent / assent.

Ages: 8 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Patients, of both sexes, affected by idiopathic scoliosis recruited at the Pediatric Orthopedics Outpatient Department of the University Hospital "Istituto di Cura Città di Pavia".
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-10-11 (Estimated); Primary Completion 2022-02-11 (Estimated); Study Completion 2022-02-11 (Estimated)

PRIMARY OUTCOMES:
Balance during self-elongation movement | 15 minutes
  To evaluate the acute effects of the self-elongation movement on the balance of patients with idiopathic scoliosis, mainly in the area of postural oscillations (oscillation area).

SECONDARY OUTCOMES:
Size of the major curve | 15 minutes
  Evaluate the acute effects of the self-elongation movement on the amplitude of the major scoliotic curve, detected with Spine 3D.
Number of patients who improve balance | 15 minutes
  Estimation of the frequency of subjects who, following self-elongation, present an improvement in balance

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marin, PhD, Principal Investigator — Laboratory of Adapted Motor Activity (LAMA), University of Pavia, Pavia, Italy; Febbi Massimiliano, PhD, Study Chair — Asomi College of Sciences, Marsa, Malta; Luisella Pedrotti, Prof, Study Director — University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No
IPD sharing will take place upon direct request and after having defined a method that fully respects the privacy of the participants

REFERENCES:
- [Background] Schreiber S, Parent EC, Moez EK, Hedden DM, Hill D, Moreau MJ, Lou E, Watkins EM, Southon SC. The effect of Schroth exercises added to the standard of care on the quality of life and muscle endurance in adolescents with idiopathic scoliosis-an assessor and statistician blinded randomized controlled trial: "SOSORT 2015 Award Winner". Scoliosis. 2015 Sep 18;10:24. doi: 10.1186/s13013-015-0048-5. eCollection 2015. PMID 26413145
- [Background] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Background] Berdishevsky H, Lebel VA, Bettany-Saltikov J, Rigo M, Lebel A, Hennes A, Romano M, Bialek M, M'hango A, Betts T, de Mauroy JC, Durmala J. Physiotherapy scoliosis-specific exercises - a comprehensive review of seven major schools. Scoliosis Spinal Disord. 2016 Aug 4;11:20. doi: 10.1186/s13013-016-0076-9. eCollection 2016. PMID 27525315
- [Background] Le Blanc R, Labelle H, Forest F, Poitras B, Rivard CH. [Possible relationship between idiopathic scoliosis and morphologic somatotypes in adolescent females]. Ann Chir. 1995;49(8):762-7. French. PMID 8561432
- [Background] Nault ML, Allard P, Hinse S, Le Blanc R, Caron O, Labelle H, Sadeghi H. Relations between standing stability and body posture parameters in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1911-7. doi: 10.1097/00007632-200209010-00018. PMID 12221357
- [Result] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499